CLINICAL TRIAL: NCT05929664
Title: Neoadjuvant REGN2810 (Cemiplimab) in Cutaneous Basal Cell Carcinoma of the Head and Neck
Brief Title: Cemiplimab for the Treatment of Locally Advanced Head and Neck Basal Cell Carcinoma Before Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2022-0944; JT 24369 (Other: JeffTrial Number)
Record Dates: First submitted 2023-02-07; First posted 2023-07-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Basal Cell Carcinoma
MeSH Terms: interventions — cemiplimab; Immunoglobulin G; Disulfides; Specimen Handling; Magnetic Resonance Spectroscopy; X-Rays; Biopsy

STUDY DESIGN:
Intervention Model Description: No Data Available
Masking Description: No Data Available
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cemiplimab) (Experimental): Patients receive cemiplimab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may transition to SOC HHI therapy. Patients undergo CT or MRI scans and collection of blood samples throughout the trial. Patients also undergo biopsies during screening and on study.
  Interventions: Biological: Cemiplimab; Procedure: Computed Tomography; Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment; Procedure: Magnetic Resonance Imaging; Procedure: Biopsy

INTERVENTIONS:
Biological: Cemiplimab — Given IV
  Other Names: 1801342-60-8; Cemiplimab RWLC; Cemiplimab-rwlc; Immunoglobulin G4; Anti-(Human Programmed Cell Death Protein 1) (Human Monoclonal REGN2810 Heavy Chain); Disulfide with Human Monoclonal REGN2810 kappa-chain; Dimer; Libtayo; REGN2810
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT SCAN; tomography
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase II trial tests how well cemiplimab works in treating basal cell carcinoma of the head and neck that has spread to nearby tissue or lymph nodes (locally advanced) before surgery (neoadjuvant). Cemiplimab is a human recombinant monoclonal IgG4 antibody that may allow the body's immune system to work against tumor cells. Giving cemiplimab before surgery may make the tumor smaller and make it easier to remove.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess treatment response of locally advanced basal cell carcinoma (BCC) of the head and neck (BCCHN) in the neoadjuvant, presurgical setting.

SECONDARY OBJECTIVES:

I. To assess functional organ preservation with neoadjuvant Cemiplimab therapy. II. To assess pathologic response. III. To assess safety of neoadjuvant therapy. IV. To assess changes in quality of life.

EXPLORATORY OBJECTIVE:

I. To assess treatment-related changes in the immune microenvironment related to functional changes in immune cell composition.

OUTLINE:

Patients receive cemiplimab intravenously (IV) over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may transition to standard of care (SOC) hedgehog inhibitor (HHI) therapy. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) scans and collection of blood samples throughout the trial. Patients also undergo biopsies during screening and on study.

Upon completion of study treatment, patients are followed up at 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, locally-advanced BCC of the head and neck requiring greater than 30% auriculectomy, rhinectomy, upper or lower lip resection, orbital exenteration (due to lid or orbital involvement), facial nerve sacrifice or Brigham and Women's stage 2b or 3 disease of head and neck

  * Tumor Specific Inclusion Criteria
  * Tumor Site: Nose; Inclusion criteria: >= 30% involvement
  * Tumor Site: Lips; Inclusion criteria: >= 30% involvement
  * Tumor Site: Ear; Inclusion criteria: >= 30% involvement
  * Tumor Site: Eyelid; Inclusion criteria: >= 50% involvement, American Joint Committee on Cancer (AJCC) stage 3
  * Tumor Site: Facial Nerve; Inclusion criteria: Clinical determination of need for sacrifice by treating surgeon
  * Tumor Site: Orbit; Inclusion criteria: Need for exenteration based on orbital or lid involvement determined by the treating surgeon
  * Tumor Site: BCC of the HN, not otherwise included in the above; Inclusion criteria: BWH T2b: 2-3 high risk factors. T3: >= 4 high risk features or bone invasion. High risk features include: >= 2 cm, poorly differentiated histology, peak nasal inspiratory (PNI) >= 0.1 mm on biopsy or gross or radiographic perineural invasion, invasion beyond subcutaneous fat
* Male or female, aged >= 18 years of age
* Performance status 0-1
* Must have a life expectancy of at least 6 months as judged by the treating physician
* Absolute neutrophil count 1500/ul or more
* Platelets 100,000/ul or more
* Hemoglobin 9 g/dl or more
* Bilirubin less than or equal to 1.5 x the upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin < 3 mg/dl)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x the upper limit of normal
* Glomerular filtration rate (GFR) greater than or equal to 40 ml/min using the Cockcroft-Gault formula or measured creatinine clearance using 24 hours urine collection
* Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]), which must also be confirmed as negative within 28 days of the start of study drugs
* Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 90 days after the last dose of study drugs. "Women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year. Men who are receiving the study medications will be instructed to adhere to contraception for 90 days after the last dose of study drugs. Men who are azoospermic do not require contraception
* Informed Consent: All subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

* Prior radiation therapy within the past 6 months for this target cancer documented by surgeon at Visit 1, Day 0 initial assessment. (Prior surgical resection to area/tumor is acceptable)
* Any history of allergy to the study drug components
* Any concurrent malignancies: exceptions include- basal cell carcinoma of the skin at another site, chronic lymphocytic leukemia, melanoma in situ, squamous cell carcinoma of the skin of a secondary location, superficial bladder cancer or in situ cervical cancer that has undergone potentially curative therapy. Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 2 years post-diagnosis
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 Grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Patients with Grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with anti-PD1 therapy may be included only after consultation with the Study Physician.
* Any Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 28 days of study drug administration., or a prior history of allogenic organ transplantation
* Any diagnosis of a significant connective tissue disorder as determined by the treating surgeon or medical team
* Patients must not be receiving any other investigational agents
* Receipt of a live attenuated vaccine within 30 days prior to the first dose of drug on trial
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Patients must not be pregnant or breastfeeding
* Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus [positive HIV 1/2 antibodies]). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc]and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Any patient with prior immunotherapy or hedge hog inhibitor (HHI) for malignancy treatment
* Any untreated metastasis(es) to the brain that may be considered active
* History of pneumonitis with the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2027-07-05 (Estimated); Study Completion 2027-07-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 6 months post surgery (up to Day 309 +/- 3 days)
  Defined by responders at surgery by clinical assessment and radiographic measurement according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Summarized by frequency counts and percentages and accompanied by exact Clopper-Pearson 95% compatibility intervals (CIs).
Disease control rate (DCR) | Up to 6 months post surgery (up to Day 309 +/- 3 days)
  Defined responders plus stable disease by clinical assessment and radiographic measurement by RECISTv1.1. Summarized by frequency counts and percentages and accompanied by exact Clopper-Pearson 95% CIs.

SECONDARY OUTCOMES:
Surgical/Clinical Benefit Rate (SBR) | At surgery (Day 129 +/- 3 days)
  Percentage of patients with an organ at risk demonstrating tumor response allowing functional organ preservation surgery.
Pathologic complete response (pCR) | Up to 6 months post surgery (up to Day 309 +/- 3 days)
  Pathologic complete response (pCR)
Major pathologic response (mPR) | Up to 6 months post surgery (up to Day 309 +/- 3 days)
  Major pathologic response (mPR)
Incidence of adverse events | Up to 6 months post surgery (up to Day 309 +/- 3 days)
  Incidence of adverse events
Changes in quality of life and functional organ preservation (FHNSI) | At baseline (Day 1) to 6 months post-surgery (up to Day 309 +/- 3 days)
  Assessed by the Functional Assessment of Cancer Therapy - Head and Neck Symptom Index (FHNSI), FACE-Questionnaire (Q), Visual Function Questionnaire (VFQ)-25 validated questionnaires. Summarized with descriptive statistics and plotted graphically (i.e., with box plots). Those data will be modeled using generalized linear modeling to account for the correlation of the longitudinal observations from the same patient.
Changes in quality of life and functional organ preservation (FACE-Q) | At baseline (Day 1)
  Assessed by the Functional Assessment of Cancer Therapy Questionnaire (FACE-Q), validated questionnaires. Score range: 0-100, generally higher scores reflect a better outcome. Summarized with descriptive statistics and plotted graphically (i.e., with box plots). Those data will be modeled using generalized linear modeling to account for the correlation of the longitudinal observations from the same patient.
Changes in quality of life and functional organ preservation (VFQ-25) | At baseline (Day 1)
  Assessed by the Visual Function Questionnaire (VFQ-25) validated questionnaires. Score range: 0-100, higher scores reflect a better outcome. Summarized with descriptive statistics and plotted graphically (i.e., with box plots). Those data will be modeled using generalized linear modeling to account for the correlation of the longitudinal observations from the same patient.
Changes in quality of life and functional organ preservation (FHNSI) | 6 months post-surgery (up to Day 309 +/- 3 days)
  Assessed by the Functional Assessment of Cancer Therapy - Head and Neck Symptom Index (FHNSI) validated questionnaires. Score range: 0-40, higher scores reflect a better outcome. Summarized with descriptive statistics and plotted graphically (i.e., with box plots). Those data will be modeled using generalized linear modeling to account for the correlation of the longitudinal observations from the same patient.
Changes in quality of life and functional organ preservation (FACE-Q) | 6 months post-surgery (up to Day 309 +/- 3 days)
  Assessed by the Functional Assessment of Cancer Therapy Questionnaire (FACE-Q), validated questionnaires. Score range: 0-100, generally higher scores reflect a better outcome. Summarized with descriptive statistics and plotted graphically (i.e., with box plots). Those data will be modeled using generalized linear modeling to account for the correlation of the longitudinal observations from the same patient.
Changes in quality of life and functional organ preservation (VFQ-25) | 6 months post-surgery (up to Day 309 +/- 3 days)
  Assessed by the Visual Function Questionnaire (VFQ-25) validated questionnaires. Score range: 0-100, higher scores reflect a better outcome. Summarized with descriptive statistics and plotted graphically (i.e., with box plots). Those data will be modeled using generalized linear modeling to account for the correlation of the longitudinal observations from the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Curry, MD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - University of Miami Health System, Miami, Florida
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee